CLINICAL TRIAL: NCT05774587
Title: Mobile Health Biometrics to Prescribe Immediate Remote Physical Activity for Enhancing Uptake to Cardiac Rehabilitation
Brief Title: Mobile Health for Cardiac Rehabilitation (Motivate-CR+)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other); North Tees and Hartlepool NHS Foundation Trust (Other); Betsi Cadwaladr University Health Board (Other Government)
Responsible Party: Principal Investigator, Helen Jones, Professor Helen Jones, Liverpool John Moores University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOTIVATE-CR+
Record Dates: First submitted 2023-02-21; First posted 2023-03-17 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Event
Keywords: Health; Rehabilitation
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Parallel assignment randomized control trial
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active control (Active Comparator): Participants will complete a 3-month cardiac rehabilitation programme supported by the onsite CR service
  Interventions: Behavioral: mHealth control group
- mHealth technology assisted exercise counselling (mHealth) (Experimental): Participants will complete a walking mHealth technology assisted exercise counselling intervention. All participants will have 4 exercise consultations with their exercise specialist. The intervention will be supported by 3 mHealth elements; 1) a wrist worn fitness watch, 2) a smartphone app for patients, and 3) a coaching website for the exercise specialist. The 3 elements will be synced, allowing data to be transferred between platforms.
  Interventions: Behavioral: mHealth technology assisted exercise counselling (mHealth)

INTERVENTIONS:
Behavioral: mHealth control group — Cardiac rehab control group
  Arms: Active control
Behavioral: mHealth technology assisted exercise counselling (mHealth) — Exercise and counselling through mHealth technology
  Arms: mHealth technology assisted exercise counselling (mHealth)

SUMMARY:
The investigators aim to conduct a feasibility study to evaluate a model where mobile health (mHealth) technology supports a remote home-based PA and counselling intervention immediately post hospital discharge to increase uptake to cardiac rehabilitation. Our overall objective is to test the feasibility of an evidence-based complex intervention prior to evaluation in a future randomized control trial (RCT)

DETAILED DESCRIPTION:
The investigators will recruit 60 participants from three cardiac rehabilitation (CR) sites: Liverpool Heart and Chest NHS Foundation Trust (n=20), University Hospitals Coventry and Warwickshire NHS Trust (n=20) and North Tees and Hartlepool Foundation Trust (n=20). The participant information sheet will be added to hospital discharge packs, participants will then be contacted by the CR team immediately post-discharge as part of routine care (within 48h at our named sites). During this contact the CR team will discuss the study information. The research fellow will then contact interested participants and consent and screening will occur via video call. Written informed consent will be captured using the eSignature solution HELLOSIGN, in line with Health Regulation Authority advice.

This is a feasibility, assessor-blind, parallel group randomized control trial (RCT). Participants will be randomized and allocated to either CR standard care (control group) or exercise counselling with mHealth + CR standard care (experimental group). Assessments will be completed twice; 1) immediately post hospital discharge, before any intervention, and 2) after CR. To minimize participant burden and ensure timely completion, outcome measures will be undertaken remotely. Participants will be mailed (guaranteed next day delivery by midday) all necessary assessment resources immediately following consent. Written and video guidance on how to complete the assessments will be provided along with online support from the research fellow.

Participants will be randomised into one of two groups:

1. CR standard care control group: Participants will follow CR standard care and have contact (e.g. telephone/virtual and/or home visit) with the CR team between discharge and beginning CR. Participants will begin structured exercise at the time provided by the CR service, the structured exercise service consists of 1-2 supervised exercise sessions per week for 12 weeks at the clinical or community centre. Exercise sessions are circuit-based, cardiovascular and strength exercise of light to moderate intensity (40-70% heart rate reserve). Participants can wear an unblinded HR monitor during structured exercise provided by the CR service. As part of the study, they will also always wear a blinded optical HR monitor. Patients can keep this kit if you wish or return it to us using a pre-paid envelope. This monitor provides no feedback to participants but provides exercise intensity and adherence data to the research team remotely. Thus, participants will wear 2 watches during CR sessions to receive feedback on HR as would be the case during standard CR, but only 1 blinded watch outside CR, wear during incidental exercise/PA, as part of the study.
2. Exercise counselling with mHealth +CR standard care experimental group: Participants will co-design a personalised and progressive home-based walking program, with support from the research fellow, that starts immediately following hospital discharge and continues as an adjunct once structured exercise CR begins. Each participant's exercise program will differ, but the aim will be to increase exercise intensity and duration throughout the programme with the goal of achieving 150-minutes of moderate intensity exercise per week, when combined with structured exercise CR sessions. To assist with the transition to independent exercise and to promote long-term adherence, participants will receive 4 virtual exercise counselling sessions. The first, held within 5 days of discharge, will be used to assess current beliefs/concerns, explore the benefits of exercise and agree on a SMART (specific, measurable, achievable, relevant and time-bound) PA plan. During this initial phase, participants will be prescribed an individualised (initial duration and intensity of sessions and rate of progression) walking plan. Once structured exercise CR has begun, a second session will be held to discuss progress and refine goals with the aim of progressing the programme. At this time, home-based sessions will be performed alongside structured exercise CR sessions to increase adherence in daily life. A third meeting will be held 1 month into CR to discuss progress. A final meeting will occur at the end of CR to review progress and strategies to maintain exercise and PA. The mHealth technology supported PA and counselling intervention, MOTIVATE, is informed by social cognitive theory. An analysis of the intervention components show MOTIVATE sessions have an emphasis on behaviour change technique categories, including "Goals and Planning," and "Feedback and Monitoring" and motivational interviewing technique processes, including "Engaging" and "Evoking" designed to promote long-term adherence to PA and exercise.

The experimental intervention will be supported by 3 mHealth elements: 1. Online coaching platform for the research fellow. Within the platform the research fellow will build the co-designed exercise programme, specifying the agreed number of sessions per week. Individual exercise sessions will be built, prescribing the duration and intensity (measured through HR) of each phase i.e., warm up, workout and cool-down. Structured exercise CR sessions will also be inserted, when CR begins, so these can be tracked. These detailed exercise sessions will then be available as pre-set sessions on the fitness tracker. Throughout the intervention the online platform will also provide the research fellow access to the participant data including; daily PA, HR during exercise, rate of perceived exertion RPE (CR-10 scale) following exercise sessions and written comments on exercise sessions. 2. Smart phone app for participants (Polar Flow). Participants will access their exercise programme and track exercise and PA achievements and provide feedback on each exercise session; including a session RPE and a written comment. 3. Wrist worn fitness tracker for participants (Polar Ignite, Polar Electro). Will act like a CR specialist on participants' wrists. The Polar Ignite fitness watch features a triaxial accelerometer and optical HR monitor. Patients can keep this kit. Participants will access pre-set exercise sessions, designed by the research fellow, on the device. The prescribed duration and intensity, via HR zones, will be displayed in real time on the watch throughout the exercise session. The watch will also provide live visual and haptic (vibration) alerts, coaching participants to execute the session as prescribed. Progress towards a personalised daily PA target will also be displayed throughout the day on the watch screen. Data from the mHealth elements, including participant comments, will be used to facilitate ongoing personalised feedback. Immediately following hospital discharge and for the 1st month of walking intervention, participants will receive text messages from the research fellow after each exercise session. For the remainder of the walking intervention (including during CR), messages will be sent weekly. Participants will be able to respond to these comments and programmes will be updated if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female
* Over 18 years old
* Post myocardial infarction (MI)
* Post percutaneous coronary intervention (PCI) patients
* Referred for CR

Exclusion Criteria:

* Unable to participate in self-management programmes because of medical care needs,
* Absolute contraindications to exercise
* Unable to operate or own mobile/smartphone devices
* Declined CR standard care
* Allergies to the watch materials
* Atrial fibrillation or other arrhythmia preventing accurate heart rate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Number of patients screened, eligible and approached | 1 year
  The percentage of patients that are screened, eligible and approached
  1. decline CR (including reasons for declining)
  2. agree to CR and
  3. consent to being part of the study
  The percentage of patients that take up standard CR and reasons for drop out; and the percentage of participants that complete outcome assessments and reasons for drop out.

SECONDARY OUTCOMES:
Device derived adherence to structured exercise | Up to 27 weeks
  Number of exercise sessions per week
Device derived duration of structured exercise | Up to 27 weeks
  Numbers of minutes completed per session
Device derived intensity of structured exercise | Up to 27 weeks
  Intensity of exercise sessions performed (% of HR reserve)
Device derived physical activity adherence (GENEActiv) | 7 days (post completion of CR programme)
  Minutes of moderate or vigorous physical activity
Change in self-reported exercise behaviour via the Behaviour Regulation in Exercise Questionnaire - 2 (BREQ-2) | Up to 27 weeks
  Behaviour regulation of exercise measured by 19 questions on a 5-point Likert scale (0-4) with 1 = not true to me and 4 = very true to me
Weight | Up to 27 weeks
  Weight (kg)
Waist circumference | Up to 27 weeks
  Waist circumference (cm)
Blood pressure | Up to 27 weeks
  Blood pressure (mmHg)
Blood lipid concentrations | Up to 27 weeks
  Blood lipid concentrations made up of HDL mmol/L, LDL mmol/L, Triglycerides mmol/L levels
Health-related quality of life | Up to 27 weeks
  MacNew heart disease questionnaire has 27 questions with 7 options as an answer, 7 being high health-related quality of life and 1 being poor health-related quality of life.
Economic data completeness | Up to 27 weeks
  Euro-Quality of life-5L questionnaire Five dimensions with five options as an answer within each one, each option is coded between 1-5 with a five digit code the outcome.
  Visual scale of 0-100 with 100 being the best state and 0 being the worse state of health participants are feeling
Patient qualitative survey on intervention acceptability | Up to 27 weeks
  Study specific questionnaire (qualitative)
Patient qualitative survey on testing acceptability | Up to 27 weeks
  Study specific questionnaire (qualitative)
Patient interview to assess intervention acceptability | Up to 27 weeks
  Patient interview
Patient interview to assess testing acceptability | Up to 27 weeks
  Patient interview
HbA1c | Up to 27 weeks
  HbA1c levels measured in mmol/mol

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool John Moores University, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share

REFERENCES:
- [Derived] Crozier A, Cocks M, Hesketh K, Miller G, Mcgregor G, Thomas L, Jones H. Mobile health biometrics to prescribe immediate remote physical activity for enhancing uptake to cardiac rehabilitation (MOTIVATE-CR+): protocol for a randomised controlled feasibility trial. BMJ Open. 2024 Feb 12;14(2):e076734. doi: 10.1136/bmjopen-2023-076734. PMID 38346877